CLINICAL TRIAL: NCT04506671
Title: A Prospective, Non-randomized, in Parallel Groups Study Evaluating the Efficacy and Safety of Percutaneous Cryoablation and Partial Nephrectomy in Localized T1b Renal Tumor
Brief Title: Percutaneous Cryoablation Versus Partial Nephrectomy for T1b Renal Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Dmitry Enikeev, MD, PhD, Deputy Director for Research, I.M. Sechenov First Moscow State Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA_vs_PN
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Renal Tumor
Keywords: Cryoablation; Renal cancer; Partial nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoablation group (Experimental): Patients with T1b renal tumor and ECOQ>20
  Interventions: Procedure: Renal biopsy; Procedure: Cryoablation
- Partial nephrectomy group (Active Comparator): Patients with T1b renal tumor
  Interventions: Procedure: Partial nephrectomy

INTERVENTIONS:
Procedure: Renal biopsy — Renal biopsy will be performed prior to the cryoablation on the basis of the center and according to the current protocols
  Arms: Cryoablation group
Procedure: Cryoablation — Cryoablation under CT guidance will be performed on the basis of the center and according to the current protocols
  Arms: Cryoablation group
Procedure: Partial nephrectomy — Partial nephrectomy will be performed on the basis of the center and according to the current protocols
  Arms: Partial nephrectomy group

SUMMARY:
The aim of our study is to assess the long-term oncological and functional outcomes of cryoablation for T1b renal tumors, as well as such important parameters as the patient's quality of life after treatment, and to compare the results with those after partial nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

•CT-confirmed renal mass > 4 to 7 cm (T1b)

Exclusion Criteria:

* Multiple renal tumors;
* Recurrence of renal tumor;
* Intolerance to iodine-containing contrast agents;
* Pregnancy;
* Patients with Bosniak 4 cysts
* Presence of other oncological diseases;
* Impossibility of organ-preserving treatment due to the proximity of the tumor to the vessels or the calyx-pelvic system
* Absence of malignant pathology based on prior biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2020-05-22 (Actual); Primary Completion 2025-05-22 (Estimated); Study Completion 2025-06-22 (Estimated)

PRIMARY OUTCOMES:
Local recurrence | 5 years
  Local recurrance will be evaluated with CT after 6 months, a year, then annually - up to 5 years after the treatment

SECONDARY OUTCOMES:
Metastatic progression | 5 years
  Presence of metastases will be evaluated with CT after 6 months, a year, then annually - up to 5 years after the treatment
Quality of life assessment: The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C-30) | 5 years
  Quality of life will be assessed using scales EORTC QLQ C-30, ranging from 1 to 100, where higher score indicating a better Quality of Life
Renal function | 5 years
  Renal function will be evaluated with eGFR
Rate of adverse events | 3 months
  Rate of intra- and postoperative adverse events will be assessed according to Clavien-Dindo grade system
Blood loss | 12 months
  Pre- and postoperative Hb level
Length of hospital stay | 1 month
  Number of days spent in hospital
Pain score | 5 years
  Pain score will be assessed using visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Urology and Reproductive Health, Sechenov University., Moscow, Russia

IPD SHARING:
Plan to Share IPD: No